CLINICAL TRIAL: NCT06941545
Title: An Assessment of Gastrointestinal Function Utilizing High Resolution Gastric Mapping, Gastroduodenal Manometry, and Gastric Emptying Testing With Assessment of Acute Response to Transcutaneous Auricular Vagal Nerve Stimulation.
Brief Title: High Resolution Gastric Mapping and Gastroduodenal Manometry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nicholas Oblizajek, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-000214
Record Dates: First submitted 2025-04-09; First posted 2025-04-23 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Dyspeptic Patients undergoing clinically indicated gastroduodenal manometry study (Experimental): First arm evaluating patients undergoing clinically indicated gastroduodenal manometry evaluation with concurrent body surface gastric mapping (BSGM), with taVNS applied during the studies.
  Interventions: Device: Alimetry; Device: tVNS; Device: Gastroduodenal Manometry
- Dyspeptic patients not undergoing GDM, tested with body surface gastric mapping alone (Experimental): Participants who have been seen in the clinical setting, having undergone other clinically indicated testing, will be recruited to undergo body surface gastric mapping (BSGM). At the end of the protocolized BSGM study the patient will undergo taVNS intervention.
  Interventions: Device: Alimetry; Device: tVNS

INTERVENTIONS:
Device: Alimetry — High resolution gastric mapping of electrical gastric activity.
Device: tVNS — Transcutaneous Auricular Vagal Nerve Stimulation, electrical stimulation to the ear.
Device: Gastroduodenal Manometry — Pressure catheter evaluating gastric and duodenal pressure profiles at rest and with certain stimuli applied
  Arms: Dyspeptic Patients undergoing clinically indicated gastroduodenal manometry study

SUMMARY:
Dyspepsia is a common problem attributed to gastric sensorimotor dysfunctions ie, delayed, or less frequently rapid gastric emptying (GE), impaired gastric accommodation, and increased gastric sensation. Therapeutic options manage symptoms, and there is no FDA approved medical therapy for dyspepsia. There is a need for better objective understanding of sensorimotor dysfunction in dyspepsia, as well as noninvasive, efficacious, safe, and inexpensive treatments for dyspepsia.

The purpose of this research is to identify disturbances and characterize phenotypes in patients with functional dyspepsia, and to assess the correlations between symptoms (during the manometry and in daily life), gastric emptying, electrical activity (BSGM), and pressure activity (manometry).

ELIGIBILITY:
Inclusion Criteria

* Symptoms consistent with functional dyspepsia as defined by the ROME IV criteria for 6 months
* Ability to perform appropriate informed consent

Exclusion Criteria

* Known cardiac arrhythmia or major ECG abnormalities, i.e. cardiac conduction disturbances (2nd or 3rd degree AV block, prolonged QTc interval (> 460 msec) or bradycardia (< 45 beats/minute)
* Conditions precluding safe use of taVNS
* Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns
* Use of opioids
* Vulnerable study population
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Antral and Duodenal Contraction Frequency | During gastrointestinal motility study (approx. 8 hours)
  Summarized as frequency (number of contractions per minute)
Gastrointestinal Antral and Duodenal Contraction Amplitude | During gastrointestinal motility study (approx. 8 hours)
  Summarized as amplitude (strength of contractions)
Gastrointestinal Antral and Duodenal Phasic Pressure Activity - Motility Index | During gastrointestinal motility study (approx. 8 hours)
  Composite measure combining frequency and amplitude for overall assessment of motility
Principal Gastric Frequency | During gastrointestinal motility study (8 hours)
  Dominant frequency of gastric waves (cycles per minute)
BMI-Adjusted Amplitude | During gastrointestinal motility study (8 hours)
  Amplitude of the gastric myoelectrical signals adjusted for body mass index
Gastric Alimetry Rhythm Index (TM) | During gastrointestinal motility study (8 hours)
  Concentration of power within the gastric frequency band over time, stability of gastric rhythm
Fed:Fasted Amplitude Ratio | During gastrointestinal motility study (8 hours)
  Ratio compares the amplitude of gastric myoelectrical activity in the fed state to the fasting state, reflecting gastric response to a meal

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas R Oblizajek, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20580984